CLINICAL TRIAL: NCT00270179
Title: A Double-Blind, Placebo-Controlled Study to Determine Whether R-huEPO Can Facilitate Presurgical Autologous Blood Donation and to Determine Its Safety for This Purpose
Brief Title: A Study to Evaluate the Effectiveness and Safety of Epoetin Alfa During the Period When One is Donating One's Own Blood Before Surgery.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005926
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Anemia
Keywords: Anemia; blood transfusion; epoetin alfa; erythropoietin; surgery; self-blood donation
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the whether epoetin alfa stimulates the bone marrow to produce red blood cells and therefore increases a patient's ability to self-donate blood prior to major surgery. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production.

DETAILED DESCRIPTION:
Major surgical procedures may require several units of blood. Blood transfusions from other people may be associated with transfusion reactions that cause fever or uncommonly, blood-borne infections. However, self-blood collections may cause anemia in a patient who will be undergoing surgery a few weeks later. Previous research with epoetin alfa suggests that it increases the rate of red blood cell production and has a beneficial effect on anemia. This randomized, double-blind, placebo-controlled 21-day study is designed to determine whether intravenous epoetin alfa will stimulate a patient's bone marrow to produce red blood cells and therefore increase a patient's ability to self-donate blood prior to major surgery for joint disease. Patients will be randomly assigned to receive either epoetin alfa 600 units per kilogram of body weight or a matching volume of placebo injected into a vein on the first study day and every 3 to 4 days thereafter for 21 days, for a total of 6 doses. The primary measures of effectiveness will be determined by the number of units of blood that can be obtained from patients during the study, the change in hemoglobin and hematocrit from pre-study to post-study, and the number of transfusions required around the time of surgery. Safety will be evaluated based on laboratory tests, vital signs, and the incidence and severity of any adverse or unusual experiences associated with drug administration. The study hypothesis is that patients treated with epoetin alfa will be able to donate more units of blood for their own surgery while receiving epoetin alfa than patients receiving placebo. Epoetin alfa 600 units per kilogram or an equal volume of placebo injected into a vein on the first day of the study, and every 3 to 4 days thereafter until day 21, for a total of 6 doses.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for major orthopedic surgery
* expected to have surgery between 25 and 35 days after starting epoetin alfa and expected to require transfusion of at least 3 units of red blood
* in good general health, with no clinically significantly abnormalities in blood and urine test values, blood clotting, or tests that check for blood in the feces
* who are not severely obese

Exclusion Criteria:

* Patients with a history of blood disease other than mild anemia or currently having a percentage of red blood cells >50% of the blood
* having the presence or history of significant diseases, especially those known to be carried in the blood, to affect the blood, or that require chemotherapy or other drugs that suppress resistance to disease or red blood cells
* having a history of seizure or uncontrolled hypertension
* having clinically significant bleeding in the stomach/intestines or elsewhere
* received a blood transfusion or received androgen therapy within 1 month prior to the start of study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Study Completion 1988-05 (Actual)

PRIMARY OUTCOMES:
Units of blood that can be obtained per patient; Change from pre-study to post-study in hemoglobin and hematocrit; Transfusions required around the time of surgery

SECONDARY OUTCOMES:
Safety (clinical laboratory tests, vital signs, incidence and severity of any adverse or unusual experiences associated with drug administration)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study to evaluate the effectiveness and safety of epoetin alfa during the period when one is donating one's own blood before surgery. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=687&filename=CR005926_CSR.pdf